CLINICAL TRIAL: NCT02392156
Title: A Global, Multicenter, Observational Study Evaluating the Impact of rFVIIIFc and rFIXFc on Patient-reported Treatment Burden and Health Economic Outcomes
Brief Title: Fc factOrs and Real-World hemophiliA Patient-ReporteD Outcomes
Acronym: FORWARD
Status: Terminated | Type: Observational
Why Stopped: Study terminated due to recruitment challenges.
Sponsor: Bioverativ Therapeutics Inc. (Industry)
Collaborators: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: 997HA401
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2018-08

CONDITIONS: Hemophilia A; Hemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B | interventions — factor VIII-Fc fusion protein; factor IX Fc fusion protein; Factor VIII

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- rFVIIIFc for hemophilia A: Administered based on the clinical judgment of the Prescribing Physician and according to the local approved drug label
  Interventions: Biological: rFVIIIFc
- non-Fc (fusion protein) replacement products for hemophilia A: Administered based on the clinical judgment of the Prescribing Physician and according to the local approved drug label
  Interventions: Biological: rFVIIIFc; Drug: non-Fc FVIII replacement products
- rFIXFc for hemophilia B: Administered based on the clinical judgment of the Prescribing Physician and according to the local approved drug label
  Interventions: Biological: rFIXFc
- non-Fc factor replacement products for hemophilia B: Administered based on the clinical judgment of the Prescribing Physician and according to the local approved drug label
  Interventions: Biological: rFIXFc; Drug: non-Fc FIX replacement products

INTERVENTIONS:
Biological: rFVIIIFc — As described in the treatment arm
  Other Names: antihemophilic factor (recombinant) Fc fusion protein; Eloctate; recombinant coagulation factor VIII Fc fusion protein; efmoroctocog alfa; BIIB031
  Groups: non-Fc (fusion protein) replacement products for hemophilia A; rFVIIIFc for hemophilia A
Biological: rFIXFc — As described in the treatment arm
  Other Names: coagulation factor IX (recombinant) Fc fusion protein; Alprolix; BIIB029
  Groups: non-Fc factor replacement products for hemophilia B; rFIXFc for hemophilia B
Drug: non-Fc FVIII replacement products — Standard plasma-derived (pd) or recombinant (r) FVIII concentrate and other traditional treatment options
  Other Names: rFVIII; pdFVIII
  Groups: non-Fc (fusion protein) replacement products for hemophilia A
Drug: non-Fc FIX replacement products — Standard plasma-derived (pd) or recombinant (r) FIX concentrate and other traditional treatment options
  Other Names: rFIX; pdFIX
  Groups: non-Fc factor replacement products for hemophilia B

SUMMARY:
The primary objective of the study is to evaluate the effectiveness of prophylactic treatment with recombinant Factor VIII Fc fusion protein (rFVIIIFc) and recombinant Factor IX Fc fusion protein (rFIXFc) therapy as assessed by patient treatment burden and health economic outcomes while maintaining disease control in males with hemophilia A or B.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a medically documented diagnosis of hemophilia A or B that is being treated prophylactically with a factor replacement product not designed to have a prolonged half-life and satisfy a therapeutic indication for rFVIIIFc/rFIXFc per the approved local label
* Have at least 50 prior exposure days (EDs) to any combination of factor replacement products
* Have documented pre-study data available that confirm fulfillment of the eligibility criteria
* Have no measurable inhibitor activity in a sample obtained within 4 weeks prior to the Baseline visit, and absence of clinical signs or symptoms of decreased response to the current factor replacement product

Key Exclusion Criteria:

* Have a diagnosis of any bleeding disorder other than hemophilia A or hemophilia B or an additional coagulation disorder(s) in addition to hemophilia A or hemophilia B
* Have a prior history of anaphylaxis associated with any factor VIII (FVIII)/ factor IX (FIX) or intravenous immunoglobin administration
* Had an inhibitor within 5 years before the Baseline visit. Note: A family history of inhibitors will not exclude the patient.
* Past or current treatment with any factor replacement product with a prolonged half-life, including an Fc product, for the treatment of hemophilia

NOTE: Other Protocol Defined Inclusion/ Exclusion Criteria May Apply.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited at various locations by prescribing physicians.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2015-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Annualized number of injections for prophylactic treatment with a Factor VIII or Factor IX replacement product | Month 2 to month 14

SECONDARY OUTCOMES:
The total annualized factor consumption (in International Units [IU] per kilogram [IU/kg]) calculated for each participant | Month 2 to month 14
Change in Treatment Satisfaction Questionnaire for Medication (TSQM) | Baseline to 14 months
  TSQM V2 is a 11-item instrument designed to measure participants' satisfaction with medication within the past 2 to 3 weeks, or since their last medication use. Treatment satisfaction is assessed through side effects, effectiveness, convenience, and global satisfaction scale domains.
Change in Hemophilia Activities List (HAL) | Baseline to 14 months
  HAL is an instrument designed to measure and quantify a participant's perceived functional ability to perform activities in daily life. The HAL consists of 42 multiple choice questions within seven domains: lying/sitting/kneeling/standing, function of legs, function of arms, use of transportation, self-care, household tasks, and leisure activities.
Change in Validated Hemophilia Regimen Treatment Adherence Scale-Prophylaxis (VERITAS-Pro) | Baseline to 14 months
  VERITAS-Pro is a 24-item questionnaire designed to measure treatment adherence through six sub-scales: Time, Dose, Plan, Remember, Skip, and Communicate. Each question is quantified on a 5-point Likert scale ("Always" to "Never") that correlates with a numeric score from 1 to 5, where higher scores indicate lower treatment adherence.
Change in Wong-Baker Faces Pain Rating Scale | Baseline to 14 months
  Wong-Baker Faces Scale is a 1-item questionnaire consisting of six facial caricatures, each depicting a different level of current perceived pain intensity, ranging from a score of 0 to 10. Higher scores indicate greater pain.
Change in Work Productivity and Impairment Questionnaire plus Classroom Impairment Questions: Hemophilia Specific (WPAI+CIQ:HS) | Baseline to 14 months
  WPAI and classroom impairment questionnaire version is a 9-item questionnaire designed to measure hemophilia-related impairment in work, school, and activity level within the past 7 days. Visual analogue scales and fill-in responses are used to compute scores for absenteeism, impairment at work/school, losses in work/school productivity, and activity impairment based on scoring algorithms and presented as impairment percentages. Higher percentages indicate greater disease-related impairment
Change in Missed planned activity and productivity | Baseline to 14 months
  The purpose of these free standing questions are to capture any missed activities due to hemophilia that are not captured in other questionnaires included in the study, especially among children and adolescents.
Change in Caregiver burden | Baseline to 14 months
  The purpose of this survey is to assess how the intensive nature of caring for a hemophilia patient affects caregiver burden, providing scores on the following scales: Emotional burden, financial burden, lifestyle, social burden, and positive emotions. This will be completed by caregivers of children and adolescents younger than 18 years of age.
Number of inpatient and outpatient healthcare visits | Baseline to 14 months
  Number of hospitalizations and number of emergency room visits or number of physician outpatient clinic visits

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Bioverativ Therapeutics Inc.
Locations (2):
- United States (2):
  - Research Site, Los Angeles, California
  - Research Site, East Lansing, Michigan